CLINICAL TRIAL: NCT02284828
Title: Effects of Eslicarbazepine Acetate (BIA 2-093) on Cognition and Psychomotor Function: Single-blind, Single-centre, Single and Multiple Dose, Fixed-order, Placebocontrolled Trial in Healthy Volunteers
Brief Title: Effects of Eslicarbazepine Acetate (BIA 2-093) on Cognition and Psychomotor Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BIA-2093-123
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Results first posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group 1 BIA 2-093 (Experimental): A single dose of oral ESL 900 mg was followed by consecutive 7-day periods of: Placebo, ESL 800 mg, and ESL 1200 mg.
  Interventions: Drug: BIA 2-093

INTERVENTIONS:
Drug: BIA 2-093
  Other Names: ESL, Eslicarbazepine acetate

SUMMARY:
Single-blind, single-centre, fixed-order study to evaluate the PD effects of a single oral dose and multiple oral doses of ESL (BIA 2-093) in healthy volunteers.

DETAILED DESCRIPTION:
Single-blind, single-centre, fixed-order study to evaluate the PD effects of a single oral dose and multiple oral doses of ESL (BIA 2-093) in healthy volunteers. A single dose of oral ESL 900 mg was followed by consecutive 7-day periods of: Placebo, ESL 800 mg, and ESL 1200 mg each given QD. The single dose was chosen to assess the ESL acute response relationship with respect to cognitive and motor skill performance, and the multiple doses were chosen to further characterize the ESL dose response relationship with respect to cognitive and motor skill performance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects, 18 to 45 years of age, inclusive
* Having completed at least high school level education (based on personal report)
* Native speakers of the English language or having learned English before 12 years of age
* Understood and provided written informed consent prior to the initiation of any protocol-specific procedures
* Body mass index (BMI) was within the range of 18 to 30 kg/m2, inclusive, with a minimum weight of at least 50 kg
* Free from any clinically significant abnormality on the basis of medical history, vital signs, physical examination, 12-lead ECG, and laboratory evaluation at Screening.
* Female subjects of childbearing potential practiced abstinence or used and were willing to continue to use a medically acceptable form of birth control for at least 1 month prior to Screening and for at least 1 month after the last study drug administration. Medically acceptable forms of contraception included intrauterine device or double-barrier. Hormone-based contraceptives methods were not acceptable, because ESL may have decreased their effectiveness. Female subjects of non-childbearing potential were amenorrheic for at least 2 years or had a hysterectomy and/or bilateral oophorectomy.
* Male subjects were required to use a double-barrier form of contraception
* Subjects who were willing and able to abide by all study requirements and restrictions

Exclusion Criteria:

* History or presence of drug or alcohol dependence (excluding nicotine and caffeine), including subjects who had ever been in a drug rehabilitation program, based on medical history
* Clinically significant abnormalities on physical examination, medical history, 12-lead ECG, vital signs, or laboratory values, as judged by the investigator or designee
* Current psychiatric illness, except nicotine and caffeine dependence. Subjects with a past history of psychiatric illness were excluded at the discretion of the investigator or designee
* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition, which in the opinion of the investigator could jeopardize the safety of the subject or the validity of the study results
* Use of a non-prescription drug within 7 days prior to the first study drug administration. Unless in the opinion of the investigator or designee, the medication received did not interfere with the study procedures or data integrity or compromise the safety of the subject
* Use of any prescription medications or natural health products (except acceptable forms of birth control and hormone replacement) within 14 days prior to the first study drug administration or throughout the study, unless in the opinion of the investigator or designee, the product did not interfere with the study procedures or data integrity or compromise the safety of the subject
* Positive serum pregnancy screen following Screening or positive urine pregnancy screen at admission and on Days -1, 9, or 16
* Positive urine drug screen (5-panel MedTox kit) at Screening, Day -1, Day 9, or Day 16.
* Positive breath alcohol test at Screening, Days -1, 9, or 16
* Female subjects who were pregnant or lactating or who were planning to become pregnant within 60 days of last study drug administration
* History of allergy or hypersensitivity to ESL, related drugs, or any of the drug excipients or other drug product components
* Positive for Hepatitis B, Hepatitis C, or HIV
* Current or pending legal charges
* Treatment with any investigational drug within 30 days prior to first drug administration
* A subject who, in the opinion of the investigator or designee, was not considered to be suitable and was unlikely to comply with the study protocol for any reason

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2007-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 BIA 2-093: A single dose of oral BIA 2-093 900 mg was followed by consecutive 7-day periods of: Placebo, ESL 800 mg, and ESL 1200 mg.
Period: Overall Study
Arm/Group | Group 1 BIA 2-093
Started | 26
Completed | 22
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Group 1 BIA 2-093
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Motor Reaction Time (MRT) (ms): Change From Baseline at Each Time Point During Acute Dosing Phase
Time Frame: -1, 3, 6, and 10 hours post-dose
Measure: Mean (Standard Deviation); unit: miliseconds
Arm/Group | Group 1 BIA 2-093
Number analyzed (Participants) | 22
miliseconds
  3 hours | 4.1 (69.22)
  6 hours | 0.7 (66.37)
  10 hours | -10.8 (52.96)

2. Primary Outcome: Motor Reaction Time (MRT) (ms): Raw Values at Each Time Point During Acute Dosing Phase
Time Frame: -1, 3, 6, and 10 hours post-dose
Measure: Mean (Standard Deviation); unit: miliseconds
Arm/Group | Group 1 BIA 2-093
Number analyzed (Participants) | 22
miliseconds
  Pre-dose | 587.0 (118.51)
  3 hours | 590.3 (89.91)
  6 hours | 588.2 (94.12)
  10 hours | 576.5 (106.46)

3. Primary Outcome: Recognition Reaction Time (RRT) (ms): Change From Baseline at Each Time Point During Acute Dosing Phase
Time Frame: -1, 3, 6, and 10 hours post-dose
Measure: Mean (Standard Deviation); unit: miliseconds
Arm/Group | Group 1 BIA 2-093
Number analyzed (Participants) | 22
miliseconds
  3 hours | -11.1 (55.23)
  6 hours | -9.2 (54.67)
  10 hours | -19.3 (51.05)

4. Primary Outcome: Recognition Reaction Time (RRT) (ms): Raw Values at Each Time Point During Acute Dosing Phase
Time Frame: -1, 3, 6, and 10 hours post-dose
Measure: Mean (Standard Deviation); unit: miliseconds
Arm/Group | Group 1 BIA 2-093
Number analyzed (Participants) | 22
miliseconds
  Pre-dose | 425.0 (81.88)
  3 hours | 414.0 (53.55)
  6 hours | 419.3 (58.70)
  10 hours | 408.0 (56.40)

5. Primary Outcome: Total Reaction Time (TRT) (ms): Raw Values at Each Time Point During Acute Dosing Phase
Time Frame: -1, 3, 6, and 10 hours post-dose
Measure: Mean (Standard Deviation); unit: miliseconds
Arm/Group | Group 1 BIA 2-093
Number analyzed (Participants) | 22
miliseconds
  Pre-dose | 1011.9 (195.12)
  3 hours | 1004.3 (134.68)
  6 hours | 1007.5 (145.70)
  10 hours | 984.5 (157.72)

6. Primary Outcome: Total Reaction Time (TRT) (ms): Change From Baseline at Each Time Point During Acute Dosing Phase
Time Frame: -1, 3, 6, and 10 hours post-dose
Measure: Mean (Standard Deviation); unit: miliseconds
Arm/Group | Group 1 BIA 2-093
Number analyzed (Participants) | 22
miliseconds
  3 hours | -7.0 (119.95)
  6 hours | -8.4 (117.00)
  10 hours | -30.0 (99.67)

ADVERSE EVENTS:
Groups:
- BIA 2-093 900 mg; BIA 2-093 800 mg; BIA 2-093 1200 mg: BIA 2-093 - ESL, Eslicarbazepine acetate
- Placebo: Placebo, PLC
Arm/Group | BIA 2-093 900 mg | Placebo | BIA 2-093 800 mg | BIA 2-093 1200 mg
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 9/26 | 13/26 | 6/26 | 7/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 2-093 900 mg (N=26) | Placebo (N=26) | BIA 2-093 800 mg (N=26) | BIA 2-093 1200 mg (N=26)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 5 | 3 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 2
Somnolence (Nervous system disorders) | 2 | 3 | 0 | 2
Erythema of eyelid (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other